## **Research Consent Form**

Official Title: The Effect of Mobile Software "Let's Move" Program Developed Based

on Transtheoretical Model on Sedentary Life Behaviors of University Students

NCT ID: not yet assigned

**Record Verification:** 14.07.2022

## **Volunteer Consent Form**

## Dear participants,

Sedentary behavior is defined as any activity that results in energy expenditure at a level of 1.5 MET (Metabolic Equivalent) or less while awake, lying or sitting. In short, a lifestyle in which physical activities are irregular or absent is called sedentary life. Recent studies have shown that sedentary lifestyle behaviors increase among young people aged 15-24. It has been shown in the literature that a sedentary lifestyle leads to physical diseases such as hypertension, diabetes, cholesterol and cancer, as well as cognitive and mental problems in later ages. In this doctoral thesis, it was aimed to evaluate the effect of the "Let's Move" mobile software program, which was developed based on the Transtheoretic Model, on changing the sedentary lifestyle behaviors of university students. Research Prof. Dr. Saime EROL and Lecturer. See. It will be conducted by Gözde ÖZDEMİR.

If you agree to participate in this research; First of all, the International Physical Activity Questionnaire will be filled. According to the results of the survey, inactive and minimally active ones will be included in the research. You will be given a smart wristband/pedometer for you to use during the research, and the computer software program "Let's Move" will be shared with you for you to download to your phones. Your body weight, height, and body fat and muscle ratios will be determined by the researcher before starting the research, after 12 weeks at the beginning of the research and after 24 weeks. You will be prompted to add the measurement results to the "Let's Move" phone app. From you through the "Let's Move" phone application; You will be asked to complete the socio-demographic characteristics questionnaire, the TTM Sedentary Life Change Stages questionnaire, and the TTM Sedentary Life Scales (Decision-Making Scale and Self-Efficacy Scale) at the 12th and 24th weeks at the beginning of the research. You will be able to see the scores you got from these scales that you filled out. In the research, presentations with educational content, videos, visual contents and warning message messages will be shared with you for three months through the "Let's Move" phone application. The smart wristbands given to you will be integrated with the program. You will be able to see your daily, weekly and alltime step counts of both yourself and other participants. In this way, your active life level will be monitored. A letter of success in the form of a certificate will be sent to the first three students with the highest number of steps in the exchange phase among the

participants. There will be an interactive messaging screen with the researcher in the program. You can share your questions and suggestions with the researcher here.

The results of the research will be used for educational and scientific purposes. Personal information will not be shared with anyone during and after the research process. The possible benefits of participating in this research are that your physical activity level will increase and you will be healthier mentally and physically. The active life suggestions in the program are activities that can be done by all healthy adults and there is no anticipated harm. However, if there is any unexpected problem in your health status, it will not be suitable for you to study. In this case, you are expected to leave the research group. You are completely free to participate in this study or not. If you want to leave at any point in the study, it will be sufficient to inform the researcher who conducted the study. However, in order not to put the researchers in a difficult situation, it would be more appropriate to inform you in advance that you will withdraw from the research. There will be no punishment, reprimand or exclusion if you do not participate or leave the study. There is no right or wrong answer to the questions asked. The points you get have nothing to do with success or failure and will not affect your school life. Participants will not take any financial responsibility for the expenses to be made for the research. No payment will be made to the participants. Participation in this research is not mandatory and is voluntary. We care about your health.

Researcher
Professor Doctor
Saime EROL

Researcher
Lecturer
Gözde Özdemir

I was informed by the researchers about the research topic. I understand the research and know what is expected of me. I agree to participate voluntarily in this research under these conditions.